CLINICAL TRIAL: NCT02265770
Title: An International Clinical Program for the Diagnosis and Treatment of Children, Adolescents and Young Adults With Ependymoma
Brief Title: An International Clinical Program for the Diagnosis and Treatment of Children With Ependymoma
Acronym: SIOP-EP-II
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIOP Ependymoma II (ET-13-002); 2013-002766-39 (EudraCT Number); VHP358 (Other: CTFG (HMA))
Record Dates: First submitted 2014-09-29; First posted 2014-10-16 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Childhood Ependymoma
MeSH Terms: conditions — Familial ependymoma | interventions — Vincristine; Etoposide; Cyclophosphamide; Cisplatin; Methotrexate; Drug Therapy; Valproic Acid; Carboplatin; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Stratum 1 arm A (Experimental): Conformal radiotherapy followed by 16 weeks of VEC + CDDP.
  Interventions: Drug: 16 weeks of VEC + CDDP; Radiation: Conformal radiotherapy
- Stratum 1 arm B (Active Comparator): Conformal radiotherapy.
  Interventions: Radiation: Conformal radiotherapy
- Stratum 2 arm A (Experimental): VEC + HD-MTX followed by conformal radiotherapy +/- boost
  Interventions: Drug: VEC + HD-MTX; Radiation: conformal radiotherapy +/- boost
- Stratum 2 arm B (Active Comparator): VEC followed by conformal radiotherapy +/- boost
  Interventions: Drug: VEC; Radiation: conformal radiotherapy +/- boost
- Stratum 3 arm A (Experimental): Chemotherapy + Valproate.
  Interventions: Drug: Chemotherapy + Valproate
- Stratum 3 arm B (Active Comparator): Chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: 16 weeks of VEC + CDDP — Days 1-36-71-106: Vincristine: 1.5 mg/m² (maximal dose 2 mg) i.v.; Days 1-3-36-38-71-73-106-108: Etoposide: 100 mg/m² infused over 60 minutes; Days 1-36-71-106: Cyclophosphamide: 3000 mg/m² in 3 divided infusions (1000 mg/m²/infusion) infused over 60 minutes; Days 22-57-92: Cisplatin: 80 mg/m² over 4 hours + Vincristine:1.5 mg/m² (maximal dose 2 mg) i.v.
  Other Names: Vincristine; Etoposide; Cyclophosphamide; Cisplatin
  Arms: Stratum 1 arm A
Drug: VEC + HD-MTX — Days 1-22-43: Vincristine: 1.5 mg/m² (maximal dose 2 mg) i.v.; Days 1-3-22-24-43-45: Etoposide: 100 mg/m² infused over 60 minutes; Days 1-22-43: Cyclophosphamide: 3000 mg/m² in 3 divided infusions (1000 mg/m²/infusion) infused over 60 minutes; Days 15-36-57: Administer methotrexate at 8000 mg/m² as a 24 hour IV infusion on days 15-36-57. 10% of the dose should be given over the first hour and 90% over the remaining 23 hours. The infusion must finish at 24 hours even if it has not been completed.
  Other Names: Vincristine; Etoposide; Cyclophosphamide; Methotrexate
  Arms: Stratum 2 arm A
Drug: Chemotherapy + Valproate — Days 1-57-113-169-225-281-337: Vincristine and Carboplatin; Days 15-71-127-183-239-295-351: Vincristine and Methotrexate; Days 29-85-141-197-253-309-365: Vincristine and Cyclophosphamide; Days 43-44-99-100-154-155-211-212-267-268-323-324-379-380: Cisplatin 2-day continuous infusion.
  Valproate: initial dose 30 mg/kg/day for two weeks in 2 divided doses (BID 15 mg/kg). Increasing weekly up to 40 - 50 - 60 mg/kg/day in 2 divided doses.
  Other Names: Vincristine; Carboplatin; Methotrexate; Cyclophosphamide; Cisplatin; Valproate
  Arms: Stratum 3 arm A
Radiation: Conformal radiotherapy — Conformal radiotherapy: 59.4Gy (children <18 months or with risk factors: 54Gy). Daily fraction 1.8 Gy, 5 fractions / week.
  Arms: Stratum 1 arm A; Stratum 1 arm B
Drug: VEC — D1: Vincristine: 1.5 mg/m² (maximal dose 2 mg) i.v.; D1-D3: Etoposide: 100 mg/m² infused over 60 minutes; D1: Cyclophosphamide: 3000 mg/m² in 3 divided infusions (1000 mg/m²/infusion) infused over 60 minutes; D22: Vincristine: 1.5 mg/m² (maximal dose 2 mg) i.v.; D22-D24: Etoposide: 100 mg/m² infused over 60 minutes; D22: Cyclophosphamide: 3000 mg/m² in 3 divided infusions (1000 mg/m²/infusion) infused over 60 minutes; D43: Vincristine: 1.5 mg/m² (maximal dose 2 mg) i.v.; D43-D45: Etoposide: 100 mg/m² infused over 60 minutes; D43: Cyclophosphamide: 3000 mg/m² in 3 divided infusions (1000 mg/m²/infusion) infused over 60 minutes
  Other Names: Vincristine; Etoposide; Cyclophosphamide
  Arms: Stratum 2 arm B
Drug: Chemotherapy — Days 1-57-113-169-225-281-337: Vincristine and Carboplatin; Days 15-71-127-183-239-295-351: Vincristine and Methotrexate; Days 29-85-141-197-253-309-365: Vincristine and Cyclophosphamide; Days 43-44-99-100-154-155-211-212-267-268-323-324-379-380: Cisplatin 2-day continuous infusion.
  Other Names: Vincristine; Carboplatin; Methotrexate; Cyclophosphamide; Cisplatin
  Arms: Stratum 3 arm B
Radiation: conformal radiotherapy +/- boost — Conformal radiotherapy: 59.4Gy (children <18 months or with risk factors: 54Gy). Daily fraction 1.8 Gy, 5 fractions / week.
  In case of persistent residue : Boost of radiation 8 Gy in 2 equivalent fractions
  Arms: Stratum 2 arm A; Stratum 2 arm B

SUMMARY:
The overall aim of this project is to improve the outcome of patients diagnosed with ependymoma by improving and harmonising the staging and the standard of care of this patient population and to improve the investigators understanding of the underlying biology thereby informing future treatment.

The program will evaluate new strategies for diagnosis (centralized reviews of pathology and imaging) and new therapeutic strategies in order to develop treatment recommendations.

Patients will be stratified into different treatment subgroups according to their age, the tumour location and the outcome of the initial surgery. Each subgroup will be studied in a specific randomised study to evaluate the proposed therapeutic strategies.

Stratum 1:

The aim of the stratum 1 is to evaluate the clinical impact of 16-week chemotherapy regimen with VEC-CDDP following surgical resection and conformal radiotherapy in terms of progression free survival in patients who are > 12 months and < 22 years at diagnosis, with completely removed intra cranial Ependymoma.

Stratum 2:

This stratum is designed as a phase II trial for patients who are > 12 months and < 22 years at diagnosis, with residual disease to investigate the possible activity of HD-MTX by giving to all patients the benefit of VEC chemotherapy whilst randomising half of patients to receive additional HD-MTX.

Patients will receive conformal radiotherapy (cRT). For patients who remain with a residual inoperable disease after induction chemotherapy and cRT, an 8 Gy boost of radiotherapy to the residual tumour will be delivered immediately after the end of the cRT.

Stratum 3 This stratum is designed as a phase II trial to evaluate the benefit of postoperative dose intense chemotherapy administered alone or in combination with valproate in children <12 months of age or those not eligible to receive radiotherapy .

DETAILED DESCRIPTION:
The Ependymoma Program is a comprehensive program to improve the accuracy of the primary diagnosis of ependymoma and explore different therapeutic strategies in children, adolescents and young adults, accordingly. This program is opened to all patients diagnosed with ependymoma below the age of 22 years.

It will include a centralised review of pre and post-operative imaging to assess the completeness of the resection.

It will also include a central review of pathology to confirm the histological diagnosis. The biological markers 1q and 6q gain, Tenascin C status, NELL2 and LAMA2, RELA-fusion and molecular subgroup by methylation array will be prospectively assessed for prospective evaluation of disease subgroups. Further biological evaluations will be coordinated within the linked BIOMECA study.

After surgery and central review of imaging and pathology, patients will be offered the opportunity to undergo second look surgery, if possible. Patients will be enrolled in one of 3 different strata according to the outcome of the initial surgical resection (residual disease vs no residual disease), their age or eligibility / suitability to receive radiotherapy. These 3 different strata correspond to 3 therapeutic strategies according to the patient status.

1. Stratum 1 is designed as a randomised phase III study for patients who have had a complete resection, with no measurable residual disease (as confirmed by centrally reviewed MRI) and are > 12 months and < 22 years at diagnosis. Those patients will be randomised to receive conformal radiotherapy followed by either 16 weeks of chemotherapy with VEC-CDDP, or observation.
2. Stratum 2 is designed as a randomised phase II study for patients who have inoperable measurable residual disease and who are > 12 months and < 22 years at diagnosis. Those patients will be randomised to two different treatment schedules of chemotherapy either with VEC or VEC+ high dose methotrexate (VEC +HD-MTX). After completion of the frontline chemotherapy, patients will be assessed for response (MRI) and will receive second look surgery when feasible. For those patients who remain unresectable with residual disease despite frontline chemotherapy and for whom second line surgery is not feasible, there will be a study of the safety of a radiotherapy boost of 8 Gy that will be administered to the residual tumour immediately after the completion of the conformal radiotherapy. Patients without evidence of residual disease after the chemotherapy and/or a second look surgery are not eligible for radiotherapy boost. All patients who have not shown progression under chemotherapy will receive, as maintenance therapy, a 16 week course of VEC -CDDP following completion of radiotherapy.
3. Stratum 3 is designed as a randomised phase II chemotherapy study in children <12 months of age or those not eligible to receive radiotherapy. These patients will be randomised to receive a dose dense chemotherapy alternating myelosuppressive and relatively non-myelosuppressive drugs at 2 weekly intervals, with or without, the addition of the histone deacetylase inhibitor, valproate.

Registry: Patients that do not fulfil the inclusion criteria of one of the interventional strata will be enrolled and followed up via an observational study which will be analysed descriptively.

ELIGIBILITY:
After Initial surgery, patients will be enrolled in one of 3 different interventional strata where they will be offered a set of therapeutic interventions based on the outcome of the intervention (no measurable residue vs residual inoperable disease), their age and/or their eligibility /suitability to receive radiotherapy.

Patients with centrally and histologically confirmed intracranial ependymoma meeting the following criteria will be enrolled into one of interventional stratum:

* Age < 22 years old at diagnosis
* Newly diagnosed intracranial ependymoma of WHO grade II-III confirmed by central pathological review
* Post-menarchal female not pregnant or nursing (breast feeding) and with a negative beta-HCG pregnancy test prior to commencing the trial
* Males and females of reproductive age and childbearing potential with effective contraception for the duration of their treatment and 6 months after the completion of their treatment
* No contraindication to the use if one of the study drugs proposed by the protocol
* Patients and/or their parents or legal guardians willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedure
* No co-existent unrelated disease at the time of study entry that would render the patient unable to receive chemotherapy
* No signs of infection.

Common inclusion criteria for Strata 1 and 2:

* Age > 12 months and < 22 years at time of study entry
* No metastasis on spinal MRI and on CSF cytology assessments
* No previous radiotherapy
* No previous chemotherapy (except steroids)
* No medical contraindication to radiotherapy and chemotherapy
* Adequate bone marrow, liver and renal functions

Specific inclusion criteria for Stratum 1:

• No residual measurable ependymoma based on the central neuroradiological review (R0-1-2)

Specific inclusion criteria for Stratum 2:

• Residual non reoperable measurable ependymoma based on the central neuroradiological review (R3-4)

Inclusion criteria for Stratum 3:

* Children younger than 12 months at time of entry to study or any children ineligible to receive radiotherapy due to age at diagnosis, tumour location or clinician / parent decision and according to national criteria
* Adequate bone marrow, liver and renal functions
* No previous chemotherapy and radiotherapy
* No contraindication to chemotherapy Patients that do not fulfill the inclusion criteria of one of the interventional strata will be enrolled and followed up into an observational study and descriptive analysis will be performed.

EXCLUSION CRITERIA for all interventional strata:

* Tumour entity other than primary intracranial ependymoma
* Primary diagnosis predating the opening of SIOP Ependymoma II
* Patients with WHO grade I ependymoma including ependymoma variants: myxopapillary ependymomas and subependymomas,patients with spinal cord location of the primary tumour
* Participation within a different trial for treatment of ependymoma
* Contraindication to one of the IMP used according to the SmPCs
* Concurrent treatment with any anti-tumour agents
* Inability to tolerate chemotherapy
* Unable to tolerate intravenous hydration
* Pre-existing mucositis, peptic ulcer, inflammatory bowel disease ascites, or pleural effusion.

Strata 1 and 2:

* Ineligible to receive radiotherapy
* Patient for whom imaging remains RX despite all effort to clarify the MRI conclusion

Stratum 3:

* Pre-existing severe hepatic and/or renal damage
* Family history of severe epilepsy
* Presence of previously undiagnosed mitochondrial disorder detected by screening as part of trial
* Elevated blood ammonium and lactate level ≥ 1.5 x upper limit of the normal

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 536 (Estimated)
Dates: Start 2015-06-02 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Gross Total Resection rate | 3 years
  Overall program, depends on the stratum (from 0.5 years to 3 years)
Progression-Free Survival | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to 4.5 years
Number of treatment responders | 15 months after final patient inclusion
  Objective response to chemotherapy is measured based on SIOP-E Neuro Imaging guidelines.

SECONDARY OUTCOMES:
Number of participants undergoing a second-look surgery | 9 months
Overall Survival | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years after the final patient inclusion
Quality of Survival | from date of randomization up to 5 years after the end of treatment
  Questionnaire
Evaluation of neuropsychological morbidity | from date of randomization up to 5 years after the end of treatment
  Scores: evaluation of processing speed (WPPSI-III, WISC-IV, WAIS-IV), verbal skills (WPPSI-III, WISC-IV, WAIS-IV), fluid intelligence (WPPSI-III / Ravens, WISC-IV / Ravens, WAIS-IV / Ravens), working memory (K-ABC / Children's Memory Scale, WISC-IV, WAIS-IV), visuo-spatial abilities (Beery-Buktenica Developmental Test of Visual-Motor Integration/Wide Range Assessment of Visual Motor Abilities - WRAVMA), regarding ability (as to national policy/WIAT-II) and motoric speed (Perdue Pegboard)
Comparison of neuroendocrine morbidity | from date of randomization up to 5 years after the end of treatment
  Weight, height and head circumference, Tanner age, early and delayed pubertal onset, blood sample analysis (evaluation of TSH, fT4, LH and FSH, oestradiol, testosterone, insulin-like growth factor 1)
Number of participants with adverse events as a measure of safety and tolerability | from date of randomization up to 5 years after the end of treatment
  Determination of short and long term safety and toxicity of frontline chemotherapy based on proportion of patients experiencing toxicity grade 3 to 4 (adverse events)
Radiotherapy-free survival rate | from date of randomization until the date of first documented progression or date of death from any cause, or radiotherapy intervention, whichever came first, up to 2.5 years after the final patient inclusion
Efficacy in each molecular sub-group | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years after the final patient inclusion
  Efficacy in each molecular subtype described in terms of Progression-Free survival and Overall Survival
Concordance between central and local radiological assessment of the efficacy of post-operative chemotherapy | 15 months after final patient inclusion
  Proportion of patients in whom the result of the central radiological review confirms the local review

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LEBLOND, MD, Principal Investigator — IHOP
Locations (40):
- Medical University of Graz-Department of Pediatrics and Adolescent Medicine, Graz, Austria
- CHR de la CITADELLE, Liège, Belgium
- University Hospital Brno, Brno, Czechia
- Aarhus University Hospital, Aarhus, Denmark
- France (26):
  - CHRU STRASBOURG - Hôpital de Hautepierre, Strasbourg, Bas-Rhin
  - AP-HM - Hôpital d'Enfants de La Timone, Marseille, Bouches-du-Rhône
  - CHU Dijon - Hôpital des Enfants, Dijon, Côte d'Or
  - CHRU BESANCON - Hôpital Jean Minjoz, Besançon, Doubs
  - CHRU BREST - Hôpital Morvan, Brest, Finistère
  - CHU de Bordeaux-Hôpital des enfants Pellegrin, Bordeaux, Gironde
  - CHU de TOULOUSE - Hôpital des Enfants, Toulouse, Haute-Garonne
  - CHRU MONTPELLIER - Hôpital Arnaud de Villeneuve, Montpellier, Herault
  - CHU de RENNES - Hôpital Sud, Rennes, Ille-et-Vilaine
  - CHRU Tours - Hôpital Clocheville, Tours, Indre-et-Loire
  - CHU GRENOBLE - Hôpital Couple-Enfant, La Tronche, Isère
  - Chu Angers, Angers, Maine-et-Loire
  - CHU REIMS - American Memorial Hospital, Reims, Marne
  - CHU NANCY - Brabois Hôpital d'Enfants, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre OSCAR LAMBRET, Lille, Nord
  - CHRU Saint-Etienne, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU Clermont- Ferrand - Hôpital Estaing, Clermont-Ferrand, Puy-de-Dôme
  - Centre LEON BERARD, Lyon, Rhône
  - CHU Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
  - CHU AMIENS-PICARDIE - Hôpital Nord, Amiens, Somme
  - CHU POITIERS - Hôpital de la Milétrie, Poitiers, Vienne
  - CHU Limoges, Limoges
  - CHU Nice - Hôpital de l'Archet 2, Nice
  - CHU La Réunion, Saint-Denis
  - Fondation Institut Curie, Paris, Île-de-France Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Our Lady's Children's Hospital, Dublin, Ireland
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
- Princess Maxima Center for pediatric oncology, Utrecht, Netherlands
- Department of Paediatric, Haukeland University Hospital, Bergen, Norway
- University Medical Center Ljubljana, Ljubljana, Slovenia
- Hospitales Universitarios Virgen Macarena y Virgen del Rocío Avda, Seville, Spain
- Skåne University Hospital, Lund, Sweden
- University Children's Hospital, Zurich, Switzerland
- Queen's Medical Centre, Nottingham, United Kingdom

REFERENCES:
- [Derived] Leblond P, Massimino M, English M, Ritzmann TA, Gandola L, Calaminus G, Thomas S, Perol D, Gautier J, Grundy RG, Frappaz D. Toward Improved Diagnosis Accuracy and Treatment of Children, Adolescents, and Young Adults With Ependymoma: The International SIOP Ependymoma II Protocol. Front Neurol. 2022 Jun 2;13:887544. doi: 10.3389/fneur.2022.887544. eCollection 2022. PMID 35720069